CLINICAL TRIAL: NCT04340336
Title: A Retrospective Multicenter Study Assessing Adult Subjects Affected With Upper and/or Lower Limb Spasticity Treated With Botulinum Neurotoxin Type A (Result Study)
Brief Title: Study Assessing Adult Subjects Affected With Upper and/or Lower Limb Spasticity Treated With Botulinum Neurotoxin Type A
Acronym: RESULT
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-IT-52120-264
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe the long term use of Botulinum Neurotoxin Type A (BoNT-A) in adult subjects affected with upper and/or lower limb spasticity who received treatment with BoNT-A for a minimum of three injections cycles at three Italian centers.

The study has a retrospective design and data relating to subjects' injections cycles occurred in the past are collected. Period of observation defined in the protocol is from 2008 to 2018, but it could change for each subject according to the number of injections cycles performed. Time frame for data collection is 12 months from study start.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged ≥18 years old at the time of the first BoNT-A injection
* Diagnosed with spasticity with any cause (excluded CP)
* Treated with a minimum of three BoNT-A treatment cycles for upper limb spasticity (ULS) and/or lower limb spasticity (LLS)
* With follow up data available in the subject's medical record
* Provision of written informed consent form, to the extent required according to applicable national local regulations for a retrospective, non-interventional study

Exclusion Criteria:

* Treatments and assessments were performed at more than one centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper and/or lower limb spasticity
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Average total dose of BoNT-A | From the baseline to the end of the study (12 months)
  Average total dose per BoNT-A type in upper and/or lower limbs (this is the average total dose injected during all sessions per BoNT-A type during the study period)
Average interval between BoNT-A injections | From the baseline to the end of the study (12 months)
  Average interval between BoNT-A injections in upper and/or lower limbs for BoNT-A overall (regardless of BoNT-A type) and per BoNT-A type

SECONDARY OUTCOMES:
Average total dose per BoNT-A type in upper limbs | From the baseline to the end of the study (12 months)
  Average total dose per BoNT-A type in upper limbs in patients treated for upper and lower limbs
Average total dose per BoNT-A type in lower limbs | From the baseline to the end of the study (12 months)
  Average total dose per BoNT-A type in lower limbs in patients treated for upper and lower limbs
Number of BoNT-A injection cycles | From the baseline to the end of the study (12 months)
Average total dose per muscle in upper limbs | From the baseline to the end of the study (12 months)
Average total dose per muscle in lower limbs | From the baseline to the end of the study (12 months)
Number of switches between BoNT-A preparations | From the baseline to the end of the study (12 months)
  Number of switches between BoNT-A preparations and reasons for switch (if known): due to no efficacy, persistent weak response in not fibrotic muscle, side effects, non-availability of the product
Reason for injection | From the baseline to the end of the study (12 months)
  Reported reason for injection at each cycle: due to medical need, scheduled visit, not recorded
Reason for interruption | From the baseline to the end of the study (12 months)
  Reported reason for BoNT-A interruptions (if applicable): side effects (excessive weakness, hematoma), no efficacy, fibrosis, contractures, long lasting clinical improvement, patients never showed up again
Occurrence of treatment discontinuation | From the baseline to the end of the study (12 months)
Global Treatment Satisfaction (GTS) | From the baseline to the end of the study (12 months)
  The qualitative subjective evaluation of patient treatment satisfaction has to be collected from medical records. The physician registered the level of satisfaction from previous treatment (very satisfied, satisfied, a little satisfied, not satisfied). A numerical value is assigned to each answer in order to obtain a numerical, subjective, GTS scale. It is a 4 point scale easy to use and to elaborate for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- Italy (3):
  - Ubaldo Del Carro, Milan
  - Marecello Esposito, Milan
  - Morena Giovannelli, Roma